CLINICAL TRIAL: NCT06705634
Title: Effects of Dry Needling of C5-C6 on Shoulder Range of Motion, Strength, Tender Points, and Blood Flow
Brief Title: How Dry Needling at the Neck Affects Shoulder Movement, Strength, Pain, and Shoulder Circulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Jace Brown, Assistant Professor of Physical Therapy, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2024-354
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dry Needling Technique; Neck Pain Musculoskeletal; Shoulder Pain; Neck Pain; Dry Needling
Keywords: neck pain; shoulder pain; muscle pain; dry needling; neck tightness; shoulder tightness
MeSH Terms: conditions — Shoulder Pain; Neck Pain; Myalgia | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Pre-Test Post-Test Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Individuals with neck-shoulder pain (Experimental): Individuals with neck-shoulder pain will receive dry needling to C5-C6 multifidus of the cervical spine.
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Dry Needling — A sterile, disposable, solid filament needle (Seirin Corp., Shizuoka, Japan) will be inserted manually into the multifidus of the C5-C6 cervical muscles. Once the needle has been inserted, the needle will be pistoned in an up and down motion within the multifidus muscle at approximately 1Hz for 10 seconds and then left in-situ for 5 minutes.

SUMMARY:
Segmental facilitation, originally proposed by Korr in the 1950s, suggests that certain spinal segments can become hyperexcitable, leading to chronic pain development. In a facilitated segment, neurons governing sensory, motor, and autonomic functions are in a state of heightened sensitivity, making them responsive to normally weak stimuli. Clinical signs include non-fatigable muscle weakness, brisk reflexes, muscle hypertonicity, tenderness upon palpation, and trophic changes like an orange-peel appearance in the affected segment's innervated areas. It's hypothesized that increased synaptic excitability in facilitated segments could cause vasoconstriction and reduced blood flow, contributing to trophic changes and muscle hypertonicity.

Manual therapies like dry needling have been shown to alleviate muscle inhibition in the extremities. Previous studies have demonstrated that mobilization of the C5-6 joint can reduce non-fatigable weakness in shoulder external rotators primarily innervated by these segments. However, the neurophysiological effects of dry needling (DN) on muscle inhibition due to a facilitated segment remain unclear. While DN has been observed to increase local tissue blood flow, its potential to mitigate the clinical signs of segmental facilitation is uncertain. While DN has been observed to increase local tissue blood flow, its potential to mitigate the clinical signs of segmental facilitation is uncertain.

Therefore, this project aims to investigate whether DN applied at a facilitated segment could normalize blood flow to its associated muscles. Specifically, this study will explore whether DN at the C5-6 level improves blood flow in the infraspinatus muscle, enhances shoulder range of motion, and influences muscle strength over time. The secondary purpose is to determine whether C5-6 DN will reduce the number of tender points in the muscles supplied by C5-6.

DETAILED DESCRIPTION:
All participants are required to attend 1 on-site visit (~ 1.25-1.5 hours) at the study site (TWU). The procedures of this research study are described in the following:

1. Administration of the Consent Form, Intake Form, and Questionnaires

   At the beginning of the on-site visit, one investigator, depending on the study site and availability of the investigators, will describe the study purpose/procedures as well as the risks/benefits associated with this study to each participant. Once the participant agrees to participate in this study, the participant will be asked to sign the written consent form. Next, the participant will complete an intake form (see below and Section 9) for their demographic information and the history of their neck-shoulder pain. Each participant also will complete 3 questionnaires: (1) Brief Pain Index (BPI), (2) Quick Disability of Arm, Shoulder, and Hand Questionnaire (QuickDASH), and (3) Central Sensitization Inventory (CSI). These forms will be delivered online via Google form, or on paper if the participant prefers. These 3 questionnaires will provide information on each participant's neck-shoulder pain, function level, and degree of central sensitization/segmental facilitation.

   The BPI (see Section 9) is a 9-item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The QuickDash is a self-report questionnaire (see Section 9) used to determine how shoulder pain affects a patient's daily life and to assess the self-rated disability of patients with shoulder pain. The CSI consists of two parts: Part A is a 25-item self-report questionnaire designed to identify patients who have symptoms that may be related to central sensitization. Part B asks patients whether they have been diagnosed with 10 central sensitization syndromes, such as fibromyalgia, whiplash, and migraine.
2. Palpation Assessment for Presence of Tenderness

   During this palpation assessment, the participants will lie prone with their arms at their sides. The investigator will palpate for tender points at the following muscle groups innervated by C5-C6 to determine eligibility: (1) Cervical paraspinals at C5-6 segment, (2) rhomboids near the spine of the scapula, (3) supraspinatus muscle belly, (4) the middle of the infraspinatus muscle belly, (5) middle deltoid. A skin marker will be used to mark these 4 sites so that the investigator can assess the same locations during the re-assessments.
3. Pre-intervention Assessments

   After gathering the subjective information and confirming the eligibility of the participant, the 3 outcome measures will be collected. The outcome measures will be collected in the following order to minimize position changes that could impact blood flow: (1) blood flow parameters in prone, (2) Shoulder range of motion (ROM), (3) Shoulder external rotation strength in supine.

   - Shoulder ROM Testing: ROM testing will be performed while the participant is lying supine with the shoulder at 90° abduction and 10° of horizontal abduction and elbow at 90°flexion. The center of rotation of the goniometer will be placed over the olecranon while one arm of the goniometer will be positioned along the length of the ulna, aligned with the ulnar styloid process. The other arm will be positioned perpendicular to the ground. For both measurements of internal and external rotation, scapular compensation will be monitored by using the thumb on the coracoid process and fingers along the spine of the scapula. Each measurement will be repeated twice with the average measurements used for data analysis.
   * Shoulder ER Strength: Shoulder external rotator strength will be tested with the subject lying supine with the involved shoulder in neutral rotation, 30° shoulder abduction, 90° elbow flexion, and full forearm pronation. The tester will hold a handheld dynamometer perpendicular to the dorsal side of the distal forearm just above the ulnar styloid process (MicroFET®2, Hoggan Scientific LLC, UT). The participant will be asked to hold that position while the tester pushes hard and attempts to break the participant's resistance. The peak force will be read directly from the handheld dynamometer. The shoulder external rotator strength will be tested twice with a minimum of a minute rest between the 2 trials. The average of the 2 trials will be used for data analysis.
   * Blood flow assessment: Each participant will remain in the same position for ultrasound imaging. The ultrasound transducer will be placed perpendicular to the infraspinous fossa to visualize arterioles or arteries of the suprascapular artery as it exits below the spine of the scapula approximately 1 inch below the acromion and to quantify the velocity of blood flow near the tender points of the infraspinatus determined by palpation during the eligibility screen. The location of the transducer will be outlined after initial placement to ensure consistent placement of the transducer between the testing sessions. The spectral Doppler waveforms will be analyzed to trace the velocities throughout the cardiac cycle. The peak systolic (PSV), end diastolic velocity (EDV), resistive index (RI) and pulsatile index (PI) will be calculated using software available on the device. On a Doppler waveform, the PSV corresponds to each "peak" within the spectral window, whereas the EDV corresponds to the point marked at the end of the cardiac cycle just prior to the systolic peak. These values will be used to calculate the RI with the formula RI = (PSV - EDV)/PSV and the PI with the formula PI = (PSV - EDV)/mean velocity, where mean velocity is the average flow velocity during the cardiac cycle. Three images will be taken, with the average used for data analysis.
4. Dry Needling Intervention

   Following the baseline testing, the PI (JB) or Co-PI (SWP) will perform the dry needling intervention. All three have more than 10 years of experience with dry needling. A sterile, disposable, solid filament needle (Seirin Corp., Shizuoka, Japan) will be inserted manually into the multifidus of C5-C6 on each side of the segment. Once the needle has been inserted, the needle will be pistoned in an up-and-down motion within the multifidus muscle at approximately 1Hz for 10 seconds. The needles will then be left in-situ for 5 minutes.

   Cadaveric and Ultrasonographic Validation of Needling Placement in the Cervical Multifidus Muscle - ScienceDirect
5. Post-intervention assessment

The 4 outcome measures will be assessed in the following order to minimize position changes: (1) blood flow parameters in the prone, (2) shoulder range of motions, (3) the number of tender points in the prone position, and then (4) Shoulder ER strength in the supine position. Shoulder ER strength will be assessed 3 times: Immediately, 15 minutes, and 30 minutes after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-65 years of age
* non-specific neck-shoulder pain (over the upper trapezius or the infraspinatus area) with an average pain ≥ 2/10 on the Numeric Pain Rating Scale (score range from 0-10, 0 = no pain, 10 = unbearable pain)
* at least one tender point in one of the 5 muscles: cervical paraspinal near C5-C6 spinal segment, rhomboids, supraspinatus, infraspinatus, and deltoid.

Exclusion Criteria:

Participants will be excluded from this study if they have a contraindication to dry needling or a medical condition affecting blood flow, including but not limited to:

* Active systemic arthritis (e.g., rheumatoid arthritis, psoriatic arthritis)
* Traumatic brain injury
* Stroke Seizures/epilepsy
* Neurological disease (e.g., multiple sclerosis, muscular dystrophy, Parkinson's, spinal cord compression)
* Acute or History of Fracture of cervical spine
* Acute or History of Fracture of the shoulder
* Circulation/vascular problems (e.g., Raynaud's)
* Cancer
* Uncontrolled diabetes/high blood sugar
* Currently pregnant
* Previous neck surgery
* Previous arthroscopic shoulder surgery in the last 5 years
* Previous shoulder arthoplasty
* Taking an anticoagulant (blood thinner)
* Allergic to ultrasound gel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Peak Systolic Velocity | Change from baseline immediately following the intervention
  On a Doppler waveform, the Peak Systolic Velocity corresponds to each "peak" within the spectral window.
End Diastolic Velocity (EDV) | Change from baseline immediately following the intervention
  End Diastolic Velocity (EDV) EDV corresponds to the point marked at the end of the cardiac cycle just prior to the systolic peak.
Resistive Index (RI) | Change from baseline immediately following the intervention
  Resistive Index is used to assess the resistance in a pulsatile vascular system. The RI is defined by the the formula RI = (PSV - EDV)/PSV.
Pulsatile Index (PI) | Change from baseline immediately following the intervention
  Pulsatility index (PI) is defined as the difference between the peak systolic flow and minimum diastolic flow velocity, divided by the mean velocity recorded throughout the cardiac cycle. It is a non-invasive method of assessing vascular resistance with the use of Doppler ultrasonography. PI is defined with the formula PI = (PSV - EDV)/mean velocity, where mean velocity is the average flow velocity during the cardiac cycle.
Shoulder Range of Motion | Change from baseline immediately following the intervention
  Shoulder range of motion of internal and external rotation is the number of degrees of motion measured using standard goniometry.
Shoulder External Rotation Strength | Change from baseline immediately following the intervention, 15 minutes after the intervention, 30 minutes after the intervention
  Shoulder external rotation strength will be measured in Newtons using a handheld dynamometer at baseline and post-intervention to assess the effect of dry needling.

SECONDARY OUTCOMES:
Number of Tender Points | Change from baseline immediately following the intervention
  The number of tender points will be assessed during palpation of muscle groups innervated by C5-C6, including the cervical paraspinals (C5-6 segment), rhomboids (near the spine of the scapula), supraspinatus muscle belly, middle of the infraspinatus muscle belly, and middle deltoid.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Woman's University T. Boone Pickens Institute of Health Sciences, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the summary data are published. Data obtained through this study may be provided to qualified researchers with academic interest in Dry Needling. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Ceballos-Laita L, Jimenez-Del-Barrio S, Marin-Zurdo J, Moreno-Calvo A, Marin-Bone J, Albarova-Corral MI, Estebanez-de-Miguel E. Effectiveness of Dry Needling Therapy on Pain, Hip Muscle Strength, and Physical Function in Patients With Hip Osteoarthritis: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 May;102(5):959-966. doi: 10.1016/j.apmr.2021.01.077. Epub 2021 Feb 7. PMID 33567336